CLINICAL TRIAL: NCT04028817
Title: Evaluation of the Concentrations of Inflammatory, Protein and Oxidative Biomarkers of Parkinson's Disease After Photobiomodulation From Sublingual Laser Application - Clinical, Randomized and Blind Test
Brief Title: Sublingual Photobiomodulation in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Daysi Tobelem, Master degree, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sublingual photobiomodulation
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Parkinson Disease
Keywords: parkinson's disease; Photobiomodulation; Inflammation; Oxidative stress
MeSH Terms: conditions — Parkinson Disease; Inflammation | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group treatment (Experimental): This group will receive laser treatment combined with low intensity exercises
  Interventions: Device: photobiomodulation
- group control (Placebo Comparator): This group will receive placebo laser treatment combined with low intensity exercises
  Interventions: Device: placebo photobiomodulation

INTERVENTIONS:
Device: photobiomodulation — the intervention will occur twice a week, 18 sessions will be performed, during the sessions will be applied sublingual laser in a single point, with wavelength of 808 nm, diameter of 0.4 cm, with irradiance of 0.8 w / cm2, for 360 s, the laser applied will be of continuous wave with energy of 36J.
  Other Names: low level laser therapy
  Arms: group treatment
Device: placebo photobiomodulation — the intervention will occur twice a week, 18 sessions will be performed, during the sessions will be applied a placebo sublingual laser for 360 s.
  Arms: group control

SUMMARY:
This study evaluates the use of photobiomodulation in the treatment of patients with Parkinson's disease. Half of participants will receive treatment with low level laser therapy and exercises in combination, while the other half will receive a placebo laser combined with exercises.

ELIGIBILITY:
Inclusion Criteria:

* patients with Parkinson's disease diagnosed with the criteria of the UK Parkinsons' Disease Society Brain Bank Clinical Diagnostic Criteria
* In the stages I to III of the disease according to Hoehn & Yahr's Parkinson's disease staging scale - modified;
* Individuals of both sexes,
* with more than 50 years
* who sign the informed consent form

Exclusion Criteria:

* patients who present some adverse event during the development of the study,
* Who have another associated neurodegenerative disease,
* Have blood dyscrasia, HIV, heart failure, hepatic or renal insufficiency, infections, neoplasias, respiratory disorders, hypophysis and hypothalamus problems.
* Who fail to understand or perform procedures correctly because of physical and mental limitations.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-10 (Estimated); Primary Completion 2021-08-10 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
10-meter walk test | 1 day
  This evaluation will be carried out from the application of the tem meter walk test. The test will be performed in a straight hall, with a line 14 meters long. The first 2 meters marked, will be provided so that the patient reaches the usual walking speed, and the last 2 meters will be provided for the patient to decelerate and stop. At the start of the test, patients will receive walking guidance at a comfortable pace.

CONTACTS AND LOCATIONS:
Locations (1):
- Daysi da Cruz Tobelem, São Paulo, Brazil